CLINICAL TRIAL: NCT01738360
Title: Phase 2a Study Evaluating the Arsenic Trioxide (ATO) in Systemic Lupus (SLE)
Brief Title: Phase 2a Study Evaluating the Arsenic Trioxide (ATO) in Systemic Lupus (SLE) (Protocol LUPSENIC)
Acronym: LUPSENIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty of inclusions and a sufficient number of relevant clinical information
Sponsor: Nantes University Hospital (Other)
Collaborators: Medsenic Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC12_0021; 2012-002259-40 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Systemic Lupus
Keywords: Arsenic trioxide; Systemic Lupus; clinically; biologically active
MeSH Terms: interventions — Arsenic Trioxide

ARMS (1):
- Arsenic trioxide (Experimental): Thirteen patients will be successively included in this study at 6 different dose levels of arsenic trioxide (0.075, 0.10, 015, 0.20, 0.25 and 0.30 mg / kg / day).
  Interventions: Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Arsenic trioxide — The study duration was 30 months (24 months recruitment + 6 months follow-up).Thirteen patients will be successively included in this study at 6 different dose levels of arsenic trioxide (0.075, 0.10, 015, 0.20, 0.25 and 0.30 mg / kg / day). The treatment should be administered by IV infusion over 2 hours of D1 to D4 (conventional hospitalization) and at D8, D11, D15, D18, D22 and D25. The protocol starts at the dose of 0.10 mg / kg / day. The stage at the dose of 0.075mg/kg/day is planned in case of toxicity with the first stage at the dose of 0.10mg/kg/day.
  The course of study is as follows :
  * Pre-inclusion between D-35 and D-15
  * Ten injections during the first month distributed as follows : conventional hospitalization from D1 to D4 (one injection per day) and daily hospitalization day for injections at D8, D11, D15, D18, D22 and D25.
  * A telephone contact between D32 and D34
  * A consultation at D40 then monthly consultation at D60, D90, D120, D150 and D180

SUMMARY:
Primary objectives :

* To investigate the safety and the tolerability of ATO by IV infusions to patients with SLE,
* To determine the maximum tolerated dose of ATO.

Secondary objectives :

* Evaluation of the clinical and biological response of the SLE to ATO,
* Time of relapse in case of positive response,
* Determination of the efficacy,
* Pharmacokinetic study of ATO.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus meeting the ACR (American College of Rheumatology) criteria, progressive either SLEDAI activity score ≥ 4, despite a corticosteroid therapy ≥ 10 mg / d associated with hydroxychloroquine (in the absence of contraindication or intolerance) and / or an immunosuppressive treatment at a stable dose,
* Insured,
* Availability for hospitalization required by the protocol (conventional and daily hospitalizations).

Exclusion Criteria:

* Inability to give their signed informed consent form,
* Performans status > 2
* QTcorrected space before treatment > 0.45 seconds
* Hemoglobin less than 11g/dL
* Neutrophils rate below 1 200 / mm3
* Platelets rate below 100 Giga / mm3
* Previous history of arrhythmia or heart rhythm disorder or other rhythm trouble by referring cardiologist
* Heart disorder (progressive pericarditis, valvular disease, ...) according to cardiologist
* Family previous history of arrhythmias
* Taking drugs that potentially prolong the QT
* Hypersensitivity to the active substance of Trisenox® or any of the excipients
* Serum potassium ≤ 4 milliequivalent / L
* Magnesemia ≤ 1,8 mg / dl
* Increase corticosteroids beyond 20 mg / day within 15 days before inclusion
* Immunosuppressive treatments, thalidomide introduced within the last 3 months
* Biotherapy (rituximab, belimumab, ...) introduced within 6 months prior to inclusion
* Pregnancy or lactation
* For women of childbearing age, men and their partner : unless effective contraception for the duration of participation in the study that is 7 months
* Creatinine clearance <50 ml / min,
* Hepatocellular insufficiency (TP <50%), and / or AST (aspartate aminotransferase) / ALT (alanine aminotransferase) / ALP (alkaline phosphatase) > 2N
* HBsAg positive, DNA detectable HbS
* Infection with HIV, HBV (hepatitis B virus) or HCV (hepatitis C virus)
* Renal or progressive central neurological impairment with possible alternative therapeutic (to be discussed with the principal investigator and scientific board meeting)
* Peripheral neuropathy
* Unweaned alcoholism
* Minor
* Patients older than 65 years
* Patient having been professionally exposed to arsenic (cleaning electronic circuits for example)
* Guardianship patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cardiac adverse events whatever grade and any adverse event of grade 3 or 4 | 30 days after the last infusion
  The definition of toxicity will be based on "Common Terminology Criteria for Adverse Events, version 4" of the U.S. Department of Health and Human Services, National Institutes of Health / National Cancer Institute.
  The investigators will consider the occurrence of a significant toxicity if at least one of the following events is observed :
  * Any symptomatic toxicity (and / or abnormality) cardiac and / or QTc prolongation > 480 msec.,
  * Apart from cardiac toxicity, toxicity of any grade 3 or 4 and irreversible toxicity (within 30 days) of any grade 1 or 2.

SECONDARY OUTCOMES:
Composite response of SLE | 30 months
  Combined clinical response using the composite response of SLE or SRI (SLE Responder Index) (SLEDAI + BILAG (British Isles Lupus Assessment Group) + PGA) : a positive response is defined by a reduction of SELENA SLEDAI of at least 4 points, no worsening ( > 0,3 point) of the physician's global assessment (PGA), no new score "A" and no more than one new score "B" about BILAG. This composite index is now the benchmark tool for evaluating therapeutic protocols in SLE.
Anti-nuclear antibodies (ANA). | 30 months
  The modification of anti-nuclear antibodies (ANA).
Anti-native DNA | 30 months
  The modification of anti-native DNA.
C3 complement | 30 monhs
  The modification of C3 complement.
C4 complement | 30 months
  The modification of C4 complement.
Sedimentation rate | 30 months
  Analysis of Sedimentation rate.
Serum creatinine | 30 months
  Analysis of serum creatinine.
Proteinuria/creatinuria ratio | 30 months
  Analysis of proteinuria/creatinuria ratio.
Serum protein electrophoresis | 30 months
  Analysis of serum protein electrophoresis.
Quantitation of immunoglobulins | 30 months
  Analysis of quantitation of immunoglobulins.
Quality of life | 30 months
  Assessment of quality of life wih questionnaires SF36 and LupusQol.
Steroids | 30 months
  Reduction of the dose of steroids throughout the study.
Immunosuppressive treatments | 30 months
  Cessation of immunosuppressive treatments.
Response time | 30 months
  Response time in case of positive response.
Time to relapse | 30 months
  Time to relapse in case of positive response.
Blood test of arsenic | D1, D2, D3, D4, D8, D11, D15, D18, D22 and D25 (before and after each infusion)
  Pharmacokinetic study of arsenic plasma with analysis of potential correlations blood rates/ toxicity and response.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed HAMIDOU, Profesor, Principal Investigator — Nantes University Hospital; Zahir AMOURA, Profesor, Study Chair — AP-HP - La Pitié-Salpétrière; Jean SIBILIA, Profesor, Study Chair — CHRU de Strasbourg; Jean-François VIALLARD, Profesor, Study Chair — University Hospital, Bordeaux; Nicolas SCHLEINITZ, Profesor, Study Chair — CHU de Marseille; Eric HACHULLA, Profesor, Study Chair — CHRU de Lille
Locations (6):
- France (6):
  - CHU de Bordeaux, Bordeaux
  - CHRU de Lille, Lille
  - CHU de Marseille, Marseille
  - Nantes University Hospital, Nantes
  - AP-HP - la Pitié-Salpétrière, Paris
  - CHRU de Strasbourg, Strasbourg

REFERENCES:
- [Derived] Hamidou M, Neel A, Poupon J, Amoura Z, Ebbo M, Sibilia J, Viallard JF, Gaborit B, Volteau C, Hardouin JB, Hachulla E, Rieger F. Safety and efficacy of low-dose intravenous arsenic trioxide in systemic lupus erythematosus: an open-label phase IIa trial (Lupsenic). Arthritis Res Ther. 2021 Mar 3;23(1):70. doi: 10.1186/s13075-021-02454-6. PMID 33658052